CLINICAL TRIAL: NCT07280416
Title: Evolution of Insomnia During the First Year in Patients Newly Diagnosed With Cancer: a Longitudinal Study and Analysis of Associated Factors.
Brief Title: Evolution of Insomnia During the First Year in Patients Newly Diagnosed With Cancer
Acronym: INDICA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH2_PANTE_INDICA_PRO; Le Puy-en-Velay Hospital (Other: Le Puy-en-Velay Hospital)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cancer; Insomnia; Pain; Depression Anxiety Disorder; Quality of Life
Keywords: cancer; insomnia; pain; Depresion Anxiety disorder; longitudinal
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have just been diagnosed with cancer.: These patients will be followed up with for one year.

SUMMARY:
The diagnosis of cancer can be a major trigger for new sleep problems, especially insomnia, in people who did not have sleep issues before. Insomnia may appear early in the care pathway and can continue over time, often interacting with other physical or emotional symptoms.

The main goal of this preliminary study is to describe how insomnia develops during the first months after a cancer diagnosis in patients who had no sleep problems at the time of diagnosis. This will be done through regular follow-up over time.

A secondary aim is to identify the factors that may contribute to the onset or persistence of insomnia, such as the cancer treatments patients receive, as well as any medical or non-medical therapies used to manage sleep difficulties.

The study will also look at whether patients who develop sleep problems are referred to psychologists trained in specific therapies for insomnia, and how well they follow and adhere to these treatments.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of metastatic or non-metastatic cancer,
* Cancer treated with intravenous chemotherapy and/or immunotherapy administered intravenously or subcutaneously,
* Age ≥ 18 years,
* Ability to read and understand French,
* Patient covered by a social security system,
* Signed informed consent.

Exclusion Criteria:

* SCI questionnaire score <16
* Diagnosed or controlled sleep disorders
* Presence of severe cognitive disorders (e.g., Alzheimer's disease) or major psychiatric disorders (e.g., psychosis), as noted in the medical record, observed at recruitment, or reported by the patient
* Patient in an emergency situation, or subject to a legal protection measure (guardianship, curatorship, or judicial protection) and unable to provide consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes adult patients (≥18 years) with a confirmed diagnosis of metastatic or non-metastatic cancer, who are scheduled to receive intravenous chemotherapy and/or immunotherapy (intravenous or subcutaneous). Eligible participants must be able to read and understand French, be covered by a social security system, and provide signed informed consent. Patients must not have pre-existing sleep disorders (SCI score ≥16) and must not have severe cognitive or major psychiatric disorders that could interfere with participation. Patients in emergency situations or under legal protection measures unable to consent are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to characterize the evolution, severity, and incidence of insomnia in patients newly diagnosed with cancer | over a 12-month period
  The primary objective of this longitudinal study is to diagnose insomnia and track its evolution and severity in patients newly diagnosed with cancer over the first year after diagnosis. Two validated questionnaires will be repeatedly administered: the Sleep Condition Indicator (SCI) and the Insomnia Severity Index (ISI). The SCI, based on DSM-5 criteria, identifies probable clinical insomnia by assessing symptom frequency, duration (difficulty falling asleep, night awakenings, early awakening), and functional impact. The ISI is a 7-item questionnaire evaluating perceived sleep difficulties over the past two weeks, including sleep initiation, maintenance, early awakening, daytime functioning, and distress. Total scores classify insomnia as absent, subclinical, moderate, or severe.

SECONDARY OUTCOMES:
The secondary objective is to characterize the sleep quality in patients newly diagnosed with cancer. | over a 12-month period
  The Pittsburgh Sleep Quality Index (PSQI) is a validated 19-item self-report questionnaire assessing overall sleep quality and identifying sleep problems. A total score ≤5 indicates good sleep, while a score >5 reflects poor sleep quality, with high sensitivity and specificity. Using the results from all study participants, the overall prevalence of sleep disturbances will be calculated.
The secondary objective is to characterize cancer-related pain in patients newly diagnosed with cancer. | over a 12-month period
  Pain perception and its impact on daily functioning will be assessed using the Brief Pain Inventory (BPI). This validated questionnaire evaluates how pain affects seven aspects of a patient's life: activity, mood, walking ability, work, relationships, sleep, and enjoyment of life.
The secondary objective is to characterize cancer-related anxiety/depression in patients newly diagnosed with cancer. | over 12-months period
  Patient anxiety and depression will be assessed using the validated Hospital Anxiety and Depression Scale (HADS). Each subscale (anxiety and depression) is scored separately: ≤7 indicates no symptoms, 8-10 suggests borderline symptoms, and ≥11 reflects definite symptoms.
The secondary objective is to characterize cancer-related quality of life in patients newly diagnosed with cancer. | over 12-months period
  The EORTC QLQ-C30 is a validated questionnaire designed to assess health-related quality of life in cancer patients, regardless of tumor site. It includes 30 items covering five functional scales (physical, role, emotional, cognitive, social), three symptom scales (fatigue, pain, nausea/vomiting), a global quality of life scale, and additional symptoms common in oncology (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). Items are rated on a 4-point Likert scale, except for global quality of life, rated 1-7. It is widely used in clinical and epidemiological studies. This questionnaire will be used to assess the cancer-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- 12 boulevard du Dr Chantemesse, Le Puy-en-Velay, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF